CLINICAL TRIAL: NCT05943613
Title: Efficacy of Intrathecal Clonidine Versus Neostigmine as Adjuvants to Bupivacaine on Postoperative Maternal and Fetal Outcomes After Elective Cesarean Section: A Randomized Double Blind Controlled Trial
Brief Title: Efficacy of Intrathecal Clonidine Versus Neostigmine as Adjuvants to Bupivacaine on Postoperative Maternal and Fetal Outcomes After Elective Cesarean Section
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Yasser Mamdouh Hassan Badawy, Assistant lecturer of anesthesia and intensive care, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: Clonidine versus Neostigmine
Record Dates: First submitted 2023-06-07; First posted 2023-07-13 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Clonidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group B (Placebo Comparator): control group : will receive 2 ml (10 mg) of intrathecal hyperbaric Bupivacaine (0.5%) and another syringe containing 1 ml of Dextrose 5%.
  Interventions: Drug: Clonidine
- Group BC (Active Comparator): will receive 2 ml (10 mg) of intrathecal hyperbaric Bupivacaine (0.5%) and another syringe containing Clonidine (30 µg) diluted in Dextrose 5% to a total volume of 1 ml.
  Interventions: Drug: Clonidine
- Group BN (Active Comparator): will receive 2 ml (10 mg) of intrathecal hyperbaric Bupivacaine (0.5%) and another syringe containing Neostigmine (10 µg) diluted in Dextrose 5% to a total volume of 1 ml.
  Interventions: Drug: Clonidine

INTERVENTIONS:
Drug: Clonidine — compare the effect of intrathecal Clonidine and Neostigmine as adjuvants to Bupivacaine in elective cesarean section

SUMMARY:
The delivery of the infant into the arms of a conscious and pain free mother is one of the most exciting and rewarding moments in medicine. Neuraxial anesthesia is now the preferred technique for lower segment cesarean sections (LSCS). Although epidural, spinal, continuous spinal, and combined spinal-epidural techniques have all been advocated, most cesarean sections are performed under single-shot spinal anesthesia.

Even when a long acting local anesthetic like bupivacaine is used, the duration of spinal anesthesia (SA) is short and higher doses of analgesics are required in the postoperative period. Therefore, achieving a subarachnoid block that provides high quality postoperative analgesia of consistently prolonged duration is an attractive goal.

DETAILED DESCRIPTION:
Opioids such as morphine, fentanyl, and sufentanil have been administered intrathecally as adjuvants to increase the duration of postoperative analgesia. Although they ensure superior quality of analgesia, they are associated with many side effects such as pruritus, nausea, vomiting, urinary retention, and especially late and unpredictable respiratory depression.

This has directed the research toward the use of newer and better local anesthetic additives for SA such as neostigmine, ketamine, midazolam, and clonidine.

Neostigmine is an anticholinesterase agent which increases the acetylcholine (Ach) concentration at the cholinergic synapse by blocking the activity of true and pseudocholinesterase enzymes. In postoperative period descending noradrenergic or cholinergic antinociceptive spinal system is activated by ongoing pain causing an increase in the release of Ach, which in the presence of neostigmine results in augmented analgesia. It has no untoward side effects such as respiratory depression, pruritus, and drowsiness as experienced with intrathecal narcotics.Clonidine is an α2-receptor agonist which has gained popularity in recent times as an adjuvant in spinal anesthesia. Analgesic effect of clonidine mediated by α2-adrenoceptors situated in the dorsal horn of spinal cord. The antinociceptive properties of clonidine indicate that it might be useful as an alternative to intrathecal opioids for postoperative analgesia, thus also avoiding the adverse effect of opioids.

Neostigmine was used in different dose ranges from 5 µg to 750 µg intrathecally but a low dose of 5 µg is sufficient to cause early onset of sensory and motor block.

On the other hand, clonidine was used in different doses from 15 µg to 450 µg, and many previous studies concluded that minimum 30 µg dose of clonidine provide a significant increase in the duration of sensory block, motor block, and spinal analgesia without increasing the incidence of side effects.

Dextrose 5% is used to make the adjuvant solutions more hyperbaric because in some studies, when hyperbaric solution of neostigmine was used, the incidence of nausea and vomiting was reduced by preventing cephalic spread of the drug to the brain stem.

Stress responses to surgical trauma and postoperative pain elicit diffuse changes in hormonal secretion such as adrenocorticotropic hormone (ACTH), cortisol and prolactin, with several deleterious metabolic and cardiovascular effects that can be prevented by effective postoperative analgesia.

Cortisol is a key player in the stress response and its secretion is facilitated by the ACTH which interacts with the sympathetic nervous system and the inhibitory control of endogenous opioid peptides, influencing pain processing.(12) Negative associations between cortisol levels and subsequent pain perception suggest the possibility that the hypothalamic-pituitary- adrenal (HPA) axis contributes to attenuating pain perception during acute stressful events, possibly mediated by increased cortisol.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ranges from 20 - 35 years old.
2. ASA physical status II.
3. Singleton fetus at term.
4. Parturient scheduled for elective lower segment cesarian section under spinal anethesia

Exclusion Criteria:

1. Patient refusal.
2. Contraindications to spinal blockade, such cardiorespiratory problems, coagulopathy, neurological disease, psychological troubles, and allergy to the used drugs.
3. Morbid obesity.
4. Failure of spinal blockade.
5. Emergency CS.
6. Complicated pregnancy.
7. Intrauterine fetal compromise.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 111 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
postoperative analgesic efficacy of intrathecal clonidine and neostigmine by use of numerical rating scale (NRS) pain score. | 2 hours after time of sensory block
  using numerical rating scale (NRS) pain score that ranges from 0 indicating no pain up to 10 indicating the worst pain

REFERENCES:
- See also: Related Info — https://www.semanticscholar.org/paper/Current-concepts-in-neuraxial-administration-of-and-Saxena-Arava/f8feed1a9cb941062de1ba8275d4928fc7c3680b
- See also: Related Info — https://link.springer.com/article/10.1007/s12630-017-0894-0
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/11374604/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/25024471/
- See also: Related Info — https://jcdr.net/article_fulltext.asp?issn=0973-709x&year=2022&month=October&volume=16&issue=10&page=UC35-UC39&id=17078